CLINICAL TRIAL: NCT04890223
Title: Efficacy of Brief Motivational Interviewing Delivered Via Mobile Instant Messaging Tools to Promote Smoking Cessation Among Unmotivated Smokers With Chronic Diseases
Brief Title: Efficacy of Brief MI Delivered Via Mobile Instant Messaging to Help Unmotivated Smokers With Chronic Diseases to Quit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NTWCREC19001_R1
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants in the intervention group will be asked to identify an unfavourable behaviour that they wish to change when filling out the baseline questionnaire. The research nurse will conduct the individual face-to-face brief MI interviews for this purpose, which will last for approximately five to ten minutes. After the face-to-face brief MI interviews, the participants in the intervention group will receive brief MI messages individually by means of mobile instant messaging for six months from the baseline. After six months, the brief MI messages will cease to be delivered to the participants in the intervention group, with whom the research team will then maintain only minimal contact until the 12-month follow-up.
  Interventions: Behavioral: Brief MI intervention
- Control group (Placebo Comparator): Participants in the control group will be asked to identify an unfavourable behaviour that they want to change at the baseline but, rather than brief MI interviews delivered face-to-face, received generic health advice consultations on the selected unfavourable behaviour that lasted approximately five to ten minutes. Each participant will receive a self-help smoking cessation booklet titled Be Smart, Quit Smoking! published by the Hong Kong Council on Smoking and Health with information about the negative health consequences of smoking, reasons to quit, strategies for quitting, and smoking cessation services available in Hong Kong along with a public quitline number (specifically, 1833183). Those who express the intention to quit at follow-ups will receive usual smoking cessation support.
  Interventions: Behavioral: Placebo intervention

INTERVENTIONS:
Behavioral: Brief MI intervention — Brief MI intervention
  Arms: Intervention group
Behavioral: Placebo intervention — Generic health advice consultations and self-help smoking cessation booklets
  Arms: Control group

SUMMARY:
This study aims to examine the efficacy of brief MI delivered by mobile instant messaging tools in promoting smoking cessation among unmotivated smokers with chronic diseases. Participants in the intervention group will receive a brief MI intervention while the control group will receive a placebo intervention.

DETAILED DESCRIPTION:
Smoking plays a causal role in the development of chronic diseases and may increase the risk of disease progression or recurrence, elevate the risk of mortality, and reduce the efficacy of treatment for disease sufferers. However, a majority of smokers with chronic diseases are unmotivated, having no intention to quit. These characteristics underscore the critical need for appropriate and effective smoking cessation interventions targeting this population. Nevertheless, most existing smoking cessation services are generic, and none seems to target smokers suffering from chronic diseases. A systematic review indicated that no study had yet examined the efficacy of a smoking cessation intervention designed specifically for unmotivated smokers with chronic diseases. Though MI was effective in promoting smoking cessation among the general population, was not effective for smokers with chronic diseases, who as has been seen tend to be unmotivated smokers. Brief MI, accordingly, is better suited to reaching these smokers in clinical settings, but the application of this approach to smoking cessation contexts has not been well studied.

The proposed intervention will be designed to promote smoking cessation among unmotivated smokers with chronic diseases. To reduce the influence of the participants' baseline characteristics on the efficacy of the intervention, this study will be designed to motivate them to change a selected unfavourable behaviour as a means to reduce their resistance to the intervention. The foot-in-the-door technique served both to facilitate the recruitment for the study and to enhance the participants' compliance with the intervention, in the latter case by promoting change in their selected unfavourable behaviour as a preliminary to further change. The rationale is that a small successful step increases readiness to take a further, larger step, in this case, smoking cessation.

Given that the exponential growth in the number of users of mobile instant messaging tools, they represent a resource for efforts to promote health and enhance treatment compliance. These were among the considerations that informed the development in this study of an intervention using brief MI delivered by mobile instant messaging tools to facilitate smoking cessation among unmotivated smokers with chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese over the age of 17
* Had smoked at least one cigarette per day over the previous three months
* Had been diagnosed with at least one chronic disease
* Able to speak Cantonese and read Chinese
* Willing to take action to improve their health but had no intention to quit smoking
* Had a smartphone and were able to use mobile instant messaging tools
* Willing to receive health promotion advice and communicate through mobile instant messaging

Exclusion Criteria:

* Participating in other smoking cessation programs or services
* With mental or cognitive impairment or communication problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Biochemically validated smoking abstinence at 12 months | 12-month follow-up
  The participants who self-reported not smoking within the past seven days will be invited to submit to a biochemical verification test of smoking abstinence, including an exhaled CO test and a salivary cotinine test. Smoking abstinence is defined as an exhaled CO level of less than 4 ppm and a saliva cotinine level lower than 15 ng/ml.

SECONDARY OUTCOMES:
Biochemically validated smoking abstinence at 6 months | 6-month follow-up
  The participants who self-reported not smoking within the past seven days will be invited to submit to a biochemical verification test of smoking abstinence, including an exhaled CO test and a salivary cotinine test. Smoking abstinence is defined as an exhaled CO level of less than 4 ppm and a saliva cotinine level lower than 15 ng/ml.
Self-reported smoking abstinence | 3-, 6-, or 12-month follow-ups
  Self-reported not smoking within the past seven days
Intention to quit | 3-, 6-, or 12-month follow-ups
  Individual's readiness to quit smoking within six months
Self-reported smoking reduction of at least 50% | 3-, 6-, or 12-month follow-ups
  Reduction in cigarette consumption from the baseline by at least 50%
Quit attempts | 3-, 6-, or 12-month follow-ups
  A period of intentional abstinence of more than 24 hours
Self-reported behavioural change | 3-, 6-, or 12-month follow-ups
  Individual's perceived modification of the selected unfavourable behaviour

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No